CLINICAL TRIAL: NCT05002530
Title: Investigating the Potential Role of Aerosolized Retinoic Acid, a Potent Vitamin A Metabolite for Treating COVID-19 Anosmia and Retinoic Acid Insufficiency .A Novel Approach for Regaining Sense of Smell.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kafrelsheikh University (Other)
Collaborators: Ministry of Health, Saudi Arabia (Other Government); The First Hospital of Jilin University (Other); Montefiore Health System and Albert Einstein College of Medicine, Newyork, United States of America (USA) (Unknown)
Responsible Party: Principal Investigator, Mahmoud Ramadan mohamed Elkazzaz, Clinical Resercher, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vitamin A and Anosmnia
Record Dates: First submitted 2021-08-10; First posted 2021-08-12 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Post COVID-19 Anosmia (Loss of Smell)
MeSH Terms: conditions — Anosmia | interventions — Vitamin D; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerosolized 13 cis retinoic acid and Vitamin D (Experimental): Patients with Post COVID-19 Anosmia (Loss of Smell) will receive one dose daily of Aerosolized 13 cis retinoic acid in gradual 2 divided doses increases from 0.2 mg/kg/day to 4 mg/kg/day as inhaled retinoic acid therapy for 3 weeks. Furthermore, the patients will receive Cholecalciferol(Vitamin D) Intramuscular injection of 600,000 units of Cholecalciferol for 2 doses given at week 0 and week 4
  Interventions: Drug: Aerosolized 13 cis retinoic acid plus Vitamin D
- Aerosolized All trans retinoic acid and Vitamin D (Experimental): Patients with Post COVID-19 Anosmia (Loss of Smell) will receive one dose daily of Aerosolized all trans retinoic acid in gradual 2 divided doses increases from 0.2 mg/kg/day to 4 mg/kg/day as inhaled retinoic acid therapy for 3 weeks. Furthermore, the patients will receive Cholecalciferol(Vitamin D) Intramuscular injection of 600,000 units of Cholecalciferol for 2 doses given at week 0 and week 4
  Interventions: Drug: Aerosolized All trans retinoic acid plus Vitamin D
- Standard therapy (Placebo Comparator): Standard therapy
  Interventions: Other: Standard therapy

INTERVENTIONS:
Drug: Aerosolized 13 cis retinoic acid plus Vitamin D — Patients with Post COVID-19 Anosmia (Loss of Smell) will receive one dose daily of Aerosolized 13 cis retinoic acid in gradual 2 divided doses increases from 0.2 mg/kg/day to 4 mg/kg/day as inhaled retinoic acid therapy for 3 weeks. Furthermore, the patients will receive Cholecalciferol(Vitamin D) Intramuscular injection of 600,000 units of Cholecalciferol for 2 doses given at week 0 and week 4
  Arms: Aerosolized 13 cis retinoic acid and Vitamin D
Drug: Aerosolized All trans retinoic acid plus Vitamin D — Patients with Post COVID-19 Anosmia (Loss of Smell) will receive one dose daily of Aerosolized All trans retinoic acid in gradual 2 divided doses increases from 0.2 mg/kg/day to 4 mg/kg/day as inhaled retinoic acid therapy for 3 weeks. Furthermore, the patients will receive Cholecalciferol(Vitamin D) Intramuscular injection of 600,000 units of Cholecalciferol for 2 doses given at week 0 and week 4
  Arms: Aerosolized All trans retinoic acid and Vitamin D
Other: Standard therapy — Standard therapy
  Arms: Standard therapy

SUMMARY:
Investigating the potential role of Aerosolized retinoic acid, a potent Vitamin A metabolite for treating COVID-19 Anosmia and retinoic acid insufficiency .A novel approach for regaining Sense of Smell.

Mahmoud ELkazzaz(1),Tamer Haydara(2), Abedelaziz Elsayed(3) ,Yousry Abo-amer(4), Hesham Attia(5), Quan Liu(6) and Amr Ahmed(7)

1. Department of chemistry and biochemistry, Faculty of Science, Damietta University, Egypt.
2. Department of Internal Medicine, Faculty of Medicine, Kafrelsheikh University, Egypt
3. Department of Pharmaceutical Biotechnology, Faculty of Pharmacy, Tanta University, Egypt.
4. Hepatology,Gastroenterology and Infectious Diseases Department, Mahala Hepatology Teaching Hospital, Egypt
5. Department of Immunology and Parasitology, Faculty of Science, Cairo University, Egypt.
6. School of Life Sciences and Engineering, Foshan University, Laboratory of Emerging Infectious Disease, Institute of Translational Medicine, The First Hospital of Jilin University, Changchun, China.
7. Director of tuberculosis program Ghubera, public health department ,First health cluster ,Ministry of health ,Saudia Arabia.

   * Very important Note: This clinical study is the first clinical study in literature (First posted August 12, 2021) which demonstrated depending on molecular findings that Vitamin A /Retinoic Acid will treat smell loss resulted by COVID-19

Recent rapidly accumulating evidences and reports indicate that partial loss of the sense of smell or even total anosmia are early markers of SARS-CoV-2 infection and frequently reported symptoms associated with the COVID-19 pandemic (Lechien J. R et al., 2020) However, the cellular mechanisms of this phenomenon are unknown. The rates of insomnia and depression were 26.45% and 9.92% in the COVID-19 patients after recovery. Therefore, finding an effective treatment for COVID-19 Anosmia is a critical point. Although, ACE2 has been identified as the principal host cell receptor of 2019-nCoV, and it is thought to play a critical role in the virus's entrance into the cell and subsequent infection, many cells can be infected by COVID-19 while also expressing little or no ACE2. Even though the COVID-19 entry receptor, angiotensin-converting enzyme 2 (ACE2), is not expressed in the receptor of olfactory neurons, or its synthesis is limited to to a minor fraction of these neurons.of these neurons, COVID-19 infection causes a loss of smell (anosmia) (Katarzyna Bilinska et al.,2021). Our recent findings showed that COVID-19 binds directly to STRA6 receptors of retinol leading to retinol depletion and retinoic acid insufficiency (M Elkazzaz et al,. 2021) . Retinoic acid insufficiency in the olfactory epithelium, both in mouse and chick models, causes progenitor cell maintenance failure and, consequently, olfactory neurons differentiation is not maintained . An explant system, showed that renewal of olfactory neurons is inhibited if retinoic acid synthesis was failed in the olfactory epithelium (Paschaki M et al., 2013) . It's worth noting that vitamin A shortage also causes olfactory and taste problems, In a study by Garrett-Laster et al., (1984), the patients had vitamin A deficiency because of malnutrition and alcoholic liver cirrhosis; they lost their sense of smell after that disorder. LaMantia and Rawson et al.,( 2007) reported that administration of retinoid acid after the damage of olfactory system motivates an immune response and produces a more quick recovery of olfactoryguided behavior. It was showed that Isotretinoin improved the significantly performance of patients in the olfactory test(Demet Kartal et al.,2017) Moreover, there is increasing evidence that retinoic acid (atRA) influences gene expression of components of renin-angiotensin system (RAS), which plays a pivotal role in the pathophysiology of essential hypertension. Retinoic acid induced ACE2 expression in different animal models. Moreover, a study suggests that topical retinoids may have applicability in promoting sinus regeneration and wound healing. In a study comparing treated and untreated nasal mucosa ,untreated regenerated mucosa showed expected changes of submucosal gland loss, basal lamina and lamina propria fibrosis and loss of cilia. Reinoic acid treatment appeared to result in better mucosal regeneration marked by less cellular atypia and fibrosis(Mendy S. Maccabee et al,. 2003).. Aerosolized retinoic acid will have an effective role in treating post COVID-19 anosmia (loss of smell) via upregulating ACE2, STRA 6 and regenerating of olfactory receptors and olfactory sensory cells and neurons.

DETAILED DESCRIPTION:
The study is a randomized interventional comparative and multicenter Phase IIII trial. 10000 adult male and female patients with post COVID-19 anosmia (loss of smell) and fulfilling the below outlined inclusion criteria will be enrolled into the study

Retinoic acids,STRA6, COVID-19, ocular and olfactory nervous system

Pinkeye (conjunctivitis), which is also associated with vitamin A deficiency, is prevalent symptom in patients with severe COVID-19 infection. (68,69).According to our findings, the binding of COVID-19 spike protein to STRA6, which is one of the main receptors for retinol cell entrance and retinoic acid production in the retina, strongly explains this symptoms .It was showed that genetic null mutation of STRA6 in mice model results in high retinoid reduction in the neurosensory retina and retinal pigment epithelium , diminished eye morphology and visual responses , despite the fact the last-mentioned problem is not as serious as in patients with mutant STRA6 (11).STRA6-mediated transport is especially significant in the eye and in the existence of vitamin A deficiency in the diet (Probable). Retinoic acid isn't transported. (70). A study strongly suggested that STRA6 works as a retinol channel/transporter(70). Analysis of function Loss- in embryos of zebrafishshowed that deficiency of Stra6 caused vitamin A deprivation of the developing eyes(70). RA signaling pathway promotes normal development of the optic nerve and ventral retina via its activities in the neural crest cell-derivedperiocular mesenchyme (71)and its deficiency may leads to retinitis. Although, several studies applied on COVID-19 patients have attempted to identify parameters linked to the olfactory disorders and taste with Angiotensin-Converting Enzyme 2 (ACE2)receptors it is clear that it takes place via receptors of vitamin A . (72) It's worth noting that vitamin A shortage also causes olfactory and taste problems, In a study by Garrett-Laster et al.,(73)the patients had vitamin A deficiency because of malnutrition and alcoholic liver cirrhosis; they lost their sense of smell after that disorder. LaMantia and Rawson reported that administration of retinoid acid after the damage of olfactory system motivates an immune response and produces a more quick recovery of olfactoryguided behavior(74).

13 cis retinoic acid improved the sense of smell and the performance of the olfactory test in acne patients (75) This also propose that insufficiency of vitamin A also rises in COVID-19.

Therefore, we strongly suggest that loss of stra6 function thorough blocking it by COVID-19 spike protein which binds to it with high affinity as a result it may hijack its signaling pathway leading to retinoic acid synthesis disruption and vitamin A deficiency . The symptoms and outcomes that arise in the eyes and nervous system of patients with COVID-19 are with unknown etiology but the results of retinoic acid deficiency manifested through vitamin A receptors. Ataxia , Headache , acute cerebrovascular disorder, impaired and consciousness are observed in patients with COVID-19 as central nervous system involvement and hyposmia, hypogeusia, neuralgia and hypopsia are seen as involvement of the peripheral nervous system. Patients with muscle involvement were also observed(76,77). COVID-19-related acute hemorrhagic necrotizing encephalopathy instances have also been documented. The unenhanced cranial BT obtained in the patients revealed hypodensity in both medial thalamuses (78). Similarly, this is a region with a lot of Stra6 receptors of Vitamin A (58). Zhao et al (79) reported the first case of Guillain-Barré syndrome linked to COVID-19.

Retinoic acids play a critical role in inducing neurogenesis and neuroplasticity. RA are important for hypothalamus and the hippocampus that control alertness and mentality .All-trans retinoic acid (atRA) can be formed from the vitamin A/ retinol in the brain. This is important for long-term potentiation (LTP). Vitamin A insufficiency also leads to circadian dysfunction. Cognitive dysfunction is also commonly showed(80,81).Pasutto et al.(7) reported that STRA6 mutations associated with lung malformations and many heart , eye diaphragm as well as retardation in mentality as in syndrome of Matthew-Wood in humans, validating its reported functions in vitamin A uptake by cells as vitamin A/retinoic acid is very critical in the process of organogenesis.

For the adult brain, components of the retinoid metabolic pathways have been thoroughly characterized(81). In some parts of the brain, all-trans-retinoic acid is synthesized.. Certain neuronal-specific genes contain recognition sequences for retinoid receptors and can be arranged directly by retinoids. receptors of retinoid have a widespread distribution in the human nervous system. This distribution differs significantly from that seen during embryonic development, implying that retinoid signalling may have a physiological role in the adult hypothalamus , cortex, striatum , amygdala, hippocampus, and other brain regions (81,82).

Retinoid signal pathways disruption in models of rodent caused in disturbance in synaptic plasticity, memory behaviors and learning . Signal pathways of retinoid also play a critical role in the pathophysiology of schizophrenia , Alzheimer's disease, and depression(81).

Retinoic acid regulates gonadotropin-releasing hormone (GnRH) and its receptor G-protein coupled receptor (GnRH) an important action in smelling process .

The olfactory bulb (OB) is a conserved region found in brain that its main function is receiving sensory neurons direct synaptic input in the nasal epithelium part and conveys that instructions to the rest of the brain. (81). It gets instructions from the brain regarding odours recognized by cells in the nasal cavity. Axons of the olfactory sensory neurons extends to the region of the olfactory bulb, which is dedicated to process odour-related instructions (82).The nervusterminalis, or zeroeth cranial nerve, contains specific neurons that produce gonadotropin-releasing hormone (GnRH). All vertebrate animals without sharks have a nervusterminalis, a chain of neurons implanted within vomeronasal or olfactory nerves in the region of the nasal canal, where it is considered a distinct nerve. The main role of the gonadotropin-releasing hormone ( GnRH) constituent of the nervusterminalis is supposed to have neuromodulatory properties . (83). Numerous studies suggested that the role of the intranasal gonadotropin-releasing hormone ( GnRH) system is to adapt and modify olfactory information, maybe at opportune times for reproduction(83). Gonadotropin-releasing hormone (GnRH), was showed to be expressed on 30 to 40 percent of neurons located in the region of the nervusterminalis and also, a small dozen of these neurons may produce gonadotropin-releasing hormone (GnRH) directly into blood veins underlying the olfactory epithelium (OE). (84). During prenatal GnRH neurons emerge from the nasal placode until reach the brain(1). These neurons become critical ingredients of the hypothalamic-pituitary-gonadal axis, which is required for activity of reproduction, after they enter the brain. Hypogonadotropichypogonadism (HH) is caused when this mechanism is disrupted (HH).

.The primary modulator of mammalian function of reproduction in both men and women is gonadotropin-releasing hormone (GnRH). It acts via distinct receptors, G-protein coupled receptor (GnRH) found in gonadotropes to induce production of the gonadotropin hormones, follicle and luteinizing -stimulating hormones (FSH), (LH)(85). a study found that congenital anosmia (loss of smell) is frequently linked with GnRH deficiency in human patients, leading to the widely held belief that GnRH neurons rely on olfactory structures to reach the brain, but this suggestion has yet to be proven(86).

Retinoic acid regulates both GnRH neurons and G-protein coupled receptor (GnRH-R).

Furthermore, retinoic acid plays critical physiological roles in synaptic plasticity, learning and memory(27), hormone production(27,28) and adult neurogenesis(27) (15).They also control a variety of processes in adults, including vision, cellular differentiation, fertilization, and tissue homeostasis(87). Retinoids are therefore essential for optimal physiology during both the early stages of development and throughout maturity(87). The mammalian type I gonadotropin releasing hormone receptor (GnRH-R) is a structurally unique G protein-coupled receptor (GPCR)(88). The majority of hormones stimulates and mediates their signal transduction via G protein-coupled receptors (GPCRs).(90) Retinoic acid induce expression of G protein-coupled receptor called Retinoic Acid - Inducible G Protein-Coupled Receptors(89) . Studies show general agreement that all-trans retinoic acid (atRA) has been linked to the regulation of G protein-coupled receptor (GPCRs) signaling,(91,92,93). Retinoic acid induces expression of G protein-coupled receptors that are used by Gonadotropin-releasing hormone (GnRH). Retinoic acid (RA) appears to be a significant regulator of GnRH neurons in GT1-1 of rat neuronal cells and hypothalamic fragments in vitro, according to a study. (93). In this study during a short period (2hours), Retinoic acid raised gonadotropin-releasing hormone (GnRH) production in a dose-dependent manner in addition, time-course tests revealed that Retinoic acid speedily induced gonadotropin-releasing hormone (GnR0H release by thirty min in both types of used cells. Furthermore, significant increase in mRNA levels of gonadotropin-releasing hormone by Retinoic acid was observed within 12hours. (94). In another study showed that that all-trans-RA controls gene expression and release of gonadotropin-releasing hormone (GnRH) in neuronal cells and hypothalamic fragments of rat. All-trans-RA increased GnRH transcription by activating functional retinoic acid response elements (RARE) in the promoter's distal region of GnRH. (95).

.

ELIGIBILITY:
Inclusion Criteria:

* adults 18 yrs or older patients
* confirmed case (+ve PCR),
* recovered/discharged (2 -ve PCR),
* suffered from sudden recent anosmia or hyposmia

Exclusion Criteria:

* Patients <18 years of age Patients who are unable to provide informed consent
* anosmia improved before COVID19 recovery,
* pregnancy
* patients who will not complete the follow up period.
* Patients without a positive COVID-19 PCR result obtained through nasopharyngeal --swab - Patients with a COVID-19 diagnosis but without self-reported anosmia --Patients with severe COVID-19 disease as defined by the Mouth Sinai Health System --Treatment Guidelines for SARS-COV-2 (requiring high flow nasal cannula, non-rebreather, CPAP/BIPAP, or mechanical ventilation OR patients requiring pressor medication OR -----
* patients with evidence of end organ damage)
* Patients with pre-existing self-reported olfactory dysfunction
* Patients with a history of chronic nasal/sinus infections (rhinosinusitis) or history of endoscopic sinus surgery
* Hypercholesterolemia
* Hypertriglyceridemia
* Patients using nasal steroid sprays or irrigations for any reason
* Patients who are prisoners of the state
* Patients who have psychiatric or developmental disorder conditions that may impair ability to provide informed consent
* Permanent blindness in one eye
* History of iritis, endophthalmitis, scleral inflammation or retinitis 15-90 days of retinal detachment or eye surgery
* The competent physician considered it inappropriate to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of olfaction | 3 weeks after beginning to take supplements
  The patient will report the degree of anosmia subjectively with score on a scale from 0 to 10 (0 means total loss of smell and 10 refers to completely normal smell sensation).

SECONDARY OUTCOMES:
Modified Brief Questionnaire of Olfactory Dysfunction (mQOD-NS) | 1 week after vitamin A softgel initiation
  The modified Brief Questionnaire of Olfactory Dysfunction - Negative Statements (QOD-NS) survey is a 17-item instrument, each item graded on a scale from 0 to 3, with total scale range from 0 to 51. Higher score indicates better olfactory-specific quality of life (QOL).
Modified Brief Questionnaire of Olfactory Dysfunction (mQOD-NS) | 2 weeks after softgel initiation
  The modified Brief Questionnaire of Olfactory Dysfunction - Negative Statements (QOD-NS) survey is a 17-item instrument, each item graded on a scale from 0 to 3, with total scale range from 0 to 51. Higher score indicates better olfactory-specific quality of life (QOL).
Modified Brief Questionnaire of Olfactory Dysfunction (mQOD-NS) | 4 weeks after softgel initiation
  The modified Brief Questionnaire of Olfactory Dysfunction - Negative Statements (QOD-NS) survey is a 17-item instrument, each item graded on a scale from 0 to 3, with total scale range from 0 to 51. Higher score indicates better olfactory-specific quality of life (QOL).
Modified Brief Questionnaire of Olfactory Dysfunction (mQOD-NS) | 6 weeks after softgel initiation
  The modified Brief Questionnaire of Olfactory Dysfunction - Negative Statements (QOD-NS) survey is a 17-item instrument, each item graded on a scale from 0 to 3, with total scale range from 0 to 51. Higher score indicates better olfactory-specific quality of life (QOL).
Sinonasal Outcomes Test | 1 week after softgel initiation
  Sino-Nasal Outcome Test (SNOT-22) is a 22-item instrument, total scale range from 0 to 110, higher score indicates more severe QOL impact.
Sinonasal Outcomes Test (SNOT-22) | 2 weeks after softgel initiation
  Sino-Nasal Outcome Test (SNOT-22) is a 22-item instrument, total scale range from 0 to 110, higher score indicates more severe QOL impact.
Sinonasal Outcomes Test (SNOT-22) | 4 weeks after softgel initiation
  Sino-Nasal Outcome Test (SNOT-22) is a 22-item instrument, total scale range from 0 to 110, higher score indicates more severe QOL impact.
Sinonasal Outcomes Test (SNOT-22) | 6 weeks after softgel initiation
  Sino-Nasal Outcome Test (SNOT-22) is a 22-item instrument, total scale range from 0 to 110, higher score indicates more severe QOL impact.
Frequency of adverse events and severe adverse events | 3 weeks
Angiotensin-converting enzyme II (ACE2) expression in lungs and olfactory region | 3 weeks
STRA6 expression in lungs and olfactory region | 3 weeks
Retinoic acid blood levels | 3 weeks
Il-6 blood levels | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tamer Haydara, Ass/Prof of Internal medicine, Study Chair — Faculty of Medicine Kafrelshiekh university; Mahmoud Elkazzaz, M.Sc of Biochemistry, Principal Investigator — Faculty of Science, Damietta university
Locations (3):
- Quan Liu, Foshan, Guangdong, China
- Tamer Haydara, Kafr ash Shaykh, Kafr Elshiekh, Egypt
- Ministry of health.First health cluster ,Riaydh, Riyadh, Saudi Arabia

REFERENCES:
- [Background] Mahmoud Elkazzaz, Tamer Haydara, Yousry Esam-Eldin Abo-Amer et al. STRA6, as A Novel Binding Receptor of COVID-19, A Breakthrough That could Explain COVID-19 Symptoms with Unknown Aetiology., 27 September 2021, PREPRINT (Version 1) available at Research Square [https://doi.org/10.21203/rs.3.rs-936697/v1]
- See also: STRA6, as A Novel Binding Receptor of COVID-19, A Breakthrough That could Explain COVID-19 Symptoms with Unknown Aetiology — https://www.researchsquare.com/article/rs-936697/v1